CLINICAL TRIAL: NCT01011049
Title: Safety and Immunogenicity of Revaccination With Influenza Vaccine in Healthy Adult Subjects Aged 18 to 64 Years Who Were Previously Vaccinated With Fluzone ID or Fluzone IM
Brief Title: Study of Influenza Vaccine Revaccination in Healthy Adults Previously Vaccinated With Fluzone ID or Fluzone IM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FID33; UTN: U1111-1111-5095 (Other: WHO)
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Fluzone Vaccine; Intradermal Injections; Adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Fluzone ID After Fluzone ID (Experimental): Participants will receive Fluzone intradermal (ID) following Fluzone ID in Study FID31
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Group 2: Fluzone IM After Fluzone ID (Experimental): Participants will receive Fluzone intramuscular (IM) following Fluzone ID in Study FID31
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Group 3: Fluzone IM After Fluzone IM (Experimental): Participants will receive Fluzone intramuscular (IM) following Fluzone IM in Study FID31
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B
- Group 4: Fluzone ID After Fluzone IM (Experimental): Participants will receive Fluzone intradermal (ID) following Fluzone intramuscular (IM) in Study FID31
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B

INTERVENTIONS:
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.1 mL, Intradermal
  Arms: Group 1: Fluzone ID After Fluzone ID
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.5 mL, Intramuscular
  Other Names: Fluzone® 2009/2010 Northern Hemisphere Formulation
  Arms: Group 2: Fluzone IM After Fluzone ID
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.5 mL, Intramuscular
  Other Names: Fluzone® 2009/2010 Northern Hemisphere Formulation
  Arms: Group 3: Fluzone IM After Fluzone IM
Biological: Influenza Virus Vaccine USP Trivalent Types A and B — 0.1 mL, Intradermal
  Arms: Group 4: Fluzone ID After Fluzone IM

SUMMARY:
The purpose of this study is to generate additional data on the immunogenicity and safety of revaccination with Fluzone Intradermal (ID) or Fluzone Intramuscular (IM) vaccine.

Primary Objective:

* To evaluate and describe the safety profile of revaccination with Fluzone ID for all participants.

Secondary Objective:

* To describe immunogenicity following revaccination with Fluzone ID or Fluzone IM.

DETAILED DESCRIPTION:
All participants, who previously received either Fluzone ID or Fluzone IM in Study FID31 (NCT 00772109), will receive one dose of either the same or the alternative vaccine.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 to 64 years on the day of vaccination in study FID33
* Enrolled in and completed study FID31 (NCT 00772109) and received the correct vaccine (Fluzone ID or Fluzone® IM) for the group to which they were randomized
* Informed consent form signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination

Exclusion Criteria :

* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* For a woman of child-bearing potential: known pregnancy or positive serum/urine pregnancy test
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the four weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period (observational trials will be allowed)
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccination in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination
* Known human immunodeficiency virus (HIV), hepatitis B surface (HBs) antigen, or Hepatitis C seropositivity.
* Previous vaccination against influenza in the past 6 months with the trial vaccine or another vaccine
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Neoplastic disease or any hematologic malignancy, (those who have localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy, as well as subjects who have a history of neoplastic disease and who have been disease free for ≥ 5 years will not be excluded).
* Personal or family history of Guillain-Barré Syndrome

Temporary Exclusion Criteria:

A prospective subject should not be included in the study until the following conditions and/or symptoms are resolved:

* Febrile illness (temperature ≥ 37.5°C [or ≥ 99.5°F]) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment
* Signs and symptoms of an acute infectious respiratory illness.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1250 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (42):
- United States (41):
  - Hoover, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Fountain Valley, California
  - San Diego, California
  - Milford, Connecticut
  - Melbourne, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Iowa City, Iowa
  - Wichita, Kansas
  - Lexington, Kentucky
  - Madisonville, Kentucky
  - Rockville, Maryland
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Endwell, New York
  - Rochester, New York
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Bensalem, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Marshfield, Wisconsin
- San Juan, Puerto Rico

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and from 23 September 2009 to 16 October 2009 in 46 medical centers in the US.
Pre-assignment Details: A total of 1248 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1: Fluzone ID After Fluzone ID: Participants who received Fluzone intradermal (ID) vaccine after receiving Fluzone ID vaccine in Study FID31 (NCT00772109)
- Group 2: Fluzone IM After Fluzone ID: Participants who received Fluzone intramuscular (IM) vaccine after receiving Fluzone intradermal (ID) vaccine in Study FID31 (NCT00772109)
- Group 3: Fluzone IM After Fluzone IM: Participants who received Fluzone intramuscular (IM) vaccine after receiving Fluzone IM vaccine in Study FID31 (NCT00772109)
- Group 4: Fluzone ID After Fluzone IM: Participants who received Fluzone intradermal (ID) vaccine after receiving Fluzone intramuscular (IM) vaccine in Study FID31 (NCT00772109)
Period: Overall Study
Arm/Group | Group 1: Fluzone ID After Fluzone ID | Group 2: Fluzone IM After Fluzone ID | Group 3: Fluzone IM After Fluzone IM | Group 4: Fluzone ID After Fluzone IM
Started | 507 | 252 | 243 | 246
Completed | 506 | 250 | 239 | 246
Not Completed | 1 | 2 | 4 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Fluzone ID After Fluzone ID | Group 2: Fluzone IM After Fluzone ID | Group 3: Fluzone IM After Fluzone IM | Group 4: Fluzone ID After Fluzone IM | Total
Number analyzed (Participants) | 507 | 252 | 243 | 246 | 1248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 507 | 252 | 242 | 246 | 1247
  >=65 years | 0 | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (13.10) | 44.8 (13.26) | 45.8 (12.74) | 43.7 (12.78) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 324 | 161 | 158 | 155 | 798
  Male | 183 | 91 | 85 | 91 | 450
Region of Enrollment [Number; unit: Participants]
  United States | 507 | 252 | 243 | 246 | 1248

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions After Vaccination With Fluzone Intradermal or Fluzone Intramuscular Vaccine
Description: Solicited injection site reactions: Erythema (redness), Swelling, Induration, Pain, Pruritus, Ecchymosis. Solicited systemic reactions: Headache, Myalgia, Malaise, Shivering, Fever (temperature).
Time Frame: Day 0 through Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1: Fluzone ID After Fluzone ID | Group 2: Fluzone IM After Fluzone ID | Group 3: Fluzone IM After Fluzone IM | Group 4: Fluzone ID After Fluzone IM
Number analyzed (Participants) | 505 | 249 | 243 | 245
Participants
  Any Solicited Injection Site Erythema | 412 | 54 | 27 | 183
  Grade 3 Erythema (≥ 5 cm) | 91 | 2 | 0 | 37
  Any Solicited Injection Site Swelling | 343 | 45 | 13 | 137
  Grade 3 Swelling (≥ 5 cm) | 40 | 4 | 2 | 14
  Any Solicited Injection Site Induration | 310 | 46 | 27 | 133
  Grade 3 Induration (≥ 5 cm) | 24 | 0 | 1 | 11
  Any Solicited Injection Site Pain | 274 | 148 | 147 | 145
  Grade 3 Pain (Incapacitating) | 5 | 4 | 2 | 2
  Any Solicited Injection Site Pruritus | 257 | 32 | 20 | 123
  Grade 3 Pruritus (Incapacitating) | 10 | 0 | 0 | 1
  Any Solicited Injection Site Ecchymosis | 53 | 10 | 10 | 25
  Grade 3 Ecchymosis (≥ 5 cm) | 1 | 0 | 1 | 0
  Any Headache | 148 | 65 | 72 | 73
  Grade 3 Headache (Prevents Daily Activities) | 13 | 4 | 3 | 5
  Any Myalgia | 131 | 77 | 75 | 68
  Grade 3 Myalgia (Prevents Daily Activities) | 8 | 5 | 0 | 7
  Any Malaise | 98 | 55 | 50 | 54
  Grade 3 Malaise (Prevents Daily Activities) | 16 | 9 | 4 | 7
  Any Shivering | 50 | 15 | 19 | 25
  Grade 3 Shivering (Prevents Daily Activities) | 8 | 0 | 0 | 5
  Any Fever | 20 | 8 | 9 | 15
  Grade 3 Fever (> 102.2 ºF) | 1 | 0 | 0 | 1

2. Secondary Outcome: Geometric Mean Titers (GMTs) Before and After Vaccination With Fluzone Intradermal or Fluzone Intramuscular Vaccine
Description: Serum antibody titers for influenza vaccine serogroups A/H1N1, A/H3N2, and B were assessed by the hemagglutinin inhibition (HAI) assay.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Serum antibody geometric mean titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Fluzone ID After Fluzone ID | Group 2: Fluzone IM After Fluzone ID | Group 3: Fluzone IM After Fluzone IM | Group 4: Fluzone ID After Fluzone IM
Number analyzed (Participants) | 495 | 242 | 234 | 240
Titers
  A/H1N1 Pre-dose (Day 0; N = 495, 242, 234, 239) | 54.5 [48.8 to 60.8] | 64.8 [55.5 to 75.7] | 51.2 [43.4 to 60.5] | 56.3 [48.7 to 65.1]
  A/H1N1 Post-dose (Day 28; N = 495, 242, 234, 239) | 142.8 [129.7 to 157.3] | 151.7 [132.1 to 174.3] | 126.2 [109.4 to 145.7] | 137.4 [119.8 to 157.5]
  A/H3N2 Pre-dose (Day 0; N = 495, 242, 234, 239) | 78.8 [69.3 to 89.5] | 91.3 [75.2 to 110.8] | 69.7 [57.9 to 84.0] | 79.7 [66.9 to 94.8]
  A/H3N2 Post-dose (Day 28; N = 495, 242, 234, 239) | 286.7 [260.3 to 315.8] | 292.0 [250.9 to 339.8] | 268.3 [234.2 to 307.3] | 290.8 [252.2 to 335.3]
  B Pre-dose (Day 0; N = 495, 242, 234, 240) | 20.1 [18.5 to 21.9] | 21.0 [18.6 to 23.6] | 21.0 [18.4 to 24.0] | 21.8 [19.3 to 24.7]
  B Post-dose (Day 28; N = 495, 242, 234, 240) | 75.0 [68.9 to 81.7] | 85.7 [75.5 to 97.3] | 73.9 [64.8 to 84.1] | 72.2 [63.1 to 82.7]

3. Secondary Outcome: Percentage of Participants Who Achieved Seroprotection Before and After Vaccination With Fluzone Intradermal or Fluzone Intramuscular Vaccine.
Description: Seroprotection was defined as a hemagglutinin inhibition (HAI) titer ≥ 1:40 at Day 28 post-vaccination.
Time Frame: Day 28 post-vaccination
Population: Serum antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Fluzone ID After Fluzone ID | Group 2: Fluzone IM After Fluzone ID | Group 3: Fluzone IM After Fluzone IM | Group 4: Fluzone ID After Fluzone IM
Number analyzed (Participants) | 495 | 242 | 234 | 240
Percentage of Participants
  A/H1N1 Pre-dose (Day 0; N = 495, 242, 234, 239) | 64 | 70 | 60 | 67
  A/H1N1 Post-dose (Day 28; N = 495, 242, 234, 239) | 92 | 94 | 92 | 90
  A/H3N2 Pre-dose (Day 0; N = 495, 242, 234, 239) | 71 | 76 | 68 | 71
  A/H3N2 Post-dose (Day 28; N = 495, 242, 234, 239) | 98 | 96 | 98 | 97
  B Pre-dose (Day 0; N = 495, 242, 234, 240) | 32 | 32 | 32 | 33
  B Post-dose (Day 28; N = 495, 242, 234, 240) | 83 | 84 | 79 | 78

4. Secondary Outcome: Percentage of Subjects Who Achieved Seroconversion After Vaccination With Fluzone Intradermal or Fluzone Intramuscular Vaccine
Description: Seroconversion was defined as either a pre vaccination hemagglutinin inhibition (HAI) titer < 1:10 and a post vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and a minimum 4 fold increase at 28 days post-vaccination.
Time Frame: Day 28 post vaccination
Population: Serum antibody titers were assessed in the per protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Fluzone ID After Fluzone ID | Group 2: Fluzone IM After Fluzone ID | Group 3: Fluzone IM After Fluzone IM | Group 4: Fluzone ID After Fluzone IM
Number analyzed (Participants) | 495 | 242 | 234 | 240
Percentage of Participants
  A/H1N1 Serogroup (N = 495, 242, 234, 239) | 31 | 29 | 26 | 30
  A/H3N2 Serogroup (N = 495, 242, 234, 239) | 47 | 40 | 42 | 44
  B Serogroup (N = 495, 242, 234, 240) | 42 | 46 | 42 | 35

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for up to 6 months, post-vaccination.
Arm/Group | Group 1: Fluzone ID After Fluzone ID | Group 2: Fluzone IM After Fluzone ID | Group 3: Fluzone IM After Fluzone IM | Group 4: Fluzone ID After Fluzone IM
Serious Adverse Events (participants affected / at risk) | 9/507 | 2/252 | 3/243 | 5/246
Other Adverse Events (participants affected / at risk) | 412/507 | 148/252 | 147/243 | 183/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Fluzone ID After Fluzone ID (N=507) | Group 2: Fluzone IM After Fluzone ID (N=252) | Group 3: Fluzone IM After Fluzone IM (N=243) | Group 4: Fluzone ID After Fluzone IM (N=246)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pituitary tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Knee arthroplasty (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal operation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: Fluzone ID After Fluzone ID (N=507) | Group 2: Fluzone IM After Fluzone ID (N=252) | Group 3: Fluzone IM After Fluzone IM (N=243) | Group 4: Fluzone ID After Fluzone IM (N=246)
Injection site erythema (General disorders) | 412/505 (412) | 54/249 (54) | 27/240 (27) | 183/245 (183)
Injection site swelling (General disorders) | 343/505 (343) | 45/249 (45) | 13/240 (13) | 137/245 (137)
Injection site induration (General disorders) | 310/505 (310) | 46/249 (46) | 27/240 (27) | 133/245 (133)
Injection site pain (Gastrointestinal disorders) | 274/505 (274) | 148/249 (148) | 147/240 (147) | 145/245 (145)
Injection site pruritus (Skin and subcutaneous tissue disorders) | 257/505 (257) | 32/249 (32) | 20/240 (20) | 123/245 (123)
Injection site ecchymosis (Vascular disorders) | 53/505 (53) | 10/249 (10) | 10/240 (10) | 25/245 (25)
Malaise (General disorders) | 98/505 (98) | 55/249 (55) | 50/240 (50) | 54/245 (54)
Shivering (General disorders) | 50/505 (50) | 15/249 (15) | 19/240 (19) | 25/245 (25)
Fever (General disorders) | 20/505 (20) | 8/249 (8) | 9/240 (9) | 15/245 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 131/505 (131) | 77/249 (77) | 75/240 (75) | 68/245 (245)
Headache (Nervous system disorders) | 148/505 (148) | 65/249 (65) | 72/240 (72) | 73/245 (73)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications